CLINICAL TRIAL: NCT06908642
Title: Evaluation of the Safety of Hemay005 Tablets in Multiple Doses and Different Administration Methods in Multiple Administrations for Chinese Adult Healthy Subjects in a Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial
Brief Title: Evaluation the Safety of hemay005 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM005CO1S01
Record Dates: First submitted 2025-03-18; First posted 2025-04-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 0-45mg Hemay005 (Active Comparator): By using titration method, the dosage of the drug was gradually increased from 0 to 45 mg BID for 14 days
  Interventions: Drug: Hemay005 tablet
- 45mg Hemay005 (Active Comparator): The subjects took the medicine twice a day, 45 mg each time, for 14 days.
  Interventions: Drug: Hemay005 tablet
- 0-60mg Hemay005 (Active Comparator): By using titration method, the dosage of the drug was gradually increased from 0 to 60 mg BID for 14 days
  Interventions: Drug: Hemay005 tablet
- 60mg Hemay005 (Active Comparator): The subjects took the medicine twice a day, 60 mg each time, for 14 days.
  Interventions: Drug: Hemay005 tablet
- 0-75 mg Hemay005 (Active Comparator): By using titration method, the dosage of the drug was gradually increased from 0 to 75 mg BID for 14 days
  Interventions: Drug: Hemay005 tablet
- 75 mg Hemay005 (Active Comparator): The subjects took the medicine twice a day, 75 mg each time, for 14 days.
  Interventions: Drug: Hemay005 tablet
- placebo (Placebo Comparator): The subjects took the medicine twice a day. In the first week, they took placebos; in the second week, they took 60 mg hemay005 each time, for a total of 14 days of medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemay005 tablet — Hemay005 is a small molecule PDE4 inhibitor.
  Arms: 0-45mg Hemay005; 0-60mg Hemay005; 0-75 mg Hemay005; 45mg Hemay005; 60mg Hemay005; 75 mg Hemay005
Drug: Placebo — Placebos are the same as drugs, but contain no Hemay005.
  Arms: placebo

SUMMARY:
Explore the influence of different administration methods (titration/non-titration) of Hemay005 tablets on the incidence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* 1) Male and female subjects aged 18 to 65 years old (inclusive of 18 and 65);
* 2) Weight: Male should be no less than 50.0 kg, female no less than 45.0 kg. Body Mass Index (BMI) [ = weight (kg) / height2 (m2) ] should be within the range of 18.5 to 30.0 kg/m2 (inclusive of boundary values);
* 3) Before the trial, they have been thoroughly informed about the nature, significance, possible benefits, as well as possible inconveniences and potential risks of the trial, and have voluntarily participated in this clinical trial. They can communicate well with the researchers, comply with all requirements of the entire study, and have signed a written informed consent form.

Exclusion Criteria:

* 1) Participants who have participated in other drug/medical device trials within the previous 3 months (based on the use of the trial drugs/medical devices);
* 2) Those with clinical manifestations of abnormalities that need to be excluded, including but not limited to diseases in the nervous system, cardiovascular system, hematological and lymphatic system, immune system, kidneys, liver, gastrointestinal tract, respiratory system, metabolism and bone system;
* 3) Those with specific allergy histories (asthma, urticaria, eczema, etc.), or with allergic constitution (such as those allergic to two or more drugs, foods or pollen), or those known to be allergic to this product;
* 4) Participants who have lost or donated blood exceeding 400ml within the previous 3 months, or those who plan to donate blood during the trial;
* 5) Pregnant or lactating women, or those who have a fertility plan or donation plan for sperm or eggs within two weeks before the trial or within 3 months after the last administration, and are unwilling or have not taken effective contraceptive measures;
* 6) General physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, hepatitis B and C, AIDS, syphilis, and HIV tests, pregnancy test for females, etc.) within the previous 7 days before randomization; electrocardiogram results within the previous 14 days before randomization judged by clinical doctors as abnormal with clinical significance; chest X-ray results within the previous 3 months before randomization judged by clinical doctors as abnormal with clinical significance;
* 7) Alcohol breath test results greater than 0.0mg/100ml or positive results in drug abuse screening;
* 8) Those who have a history of severe vomiting or diarrhea within the previous 7 days or any other diseases or physiological conditions that may interfere with the test results;
* 9) Those who have suffered from major clinical diseases or undergone major surgical operations within 3 months before screening;
* 10) Those who consume more than 14 units of alcohol per week (1 unit = 17.7 mL ethanol, which is equivalent to 357 mL of 5% alcohol beverage, 43 mL of 40% alcohol liquor, or 147 mL of 12% wine) within 3 months before screening, or those who cannot abstain from alcohol during the test;
* 11) Those who smoke more than 5 cigarettes per day on average within 3 months before screening, or those who cannot stop using any tobacco products during the test;
* 12) Those who consume excessive tea, coffee and/or beverages rich in caffeine (more than 8 cups, 1 cup = 250 mL) every day within 3 months before screening.
* 13) Exclude those who have used any drugs that inhibit or induce liver drug-metabolizing enzymes within the past 30 days (such as inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids; inhibitors - SSRI class antidepressants, cimetidine, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines).
* 14) Those with a history of tuberculosis or those with active tuberculosis during the screening period;
* 15) Those who are unable to eat or have difficulty swallowing;
* 16) Those who have used any prescription drugs, over-the-counter drugs, health supplements, herbal products or vaccines within 14 days before randomization or have stopped taking them for less than 5 half-lives;
* 17) Those who have used Apremilast or Hemay005 tablets in the past;
* 18) Those who cannot tolerate venipuncture and/or have a history of fainting or needle shock;
* 19) Those who have used any drugs within one year before screening;
* 20) Those who, in the researcher's opinion, have poor compliance or any factors that make them unsuitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Explore the influence of different administration methods (titration/non-titration) of Hemay005 tablets on the incidence of adverse reactions. | 14 Days
  Number of Participants With Treatment-Related Adverse Events as Assessed by Grade of Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China